CLINICAL TRIAL: NCT01681953
Title: A Multi-Center, Double-Blind, Randomized, Placebo-Controlled, Parallel Group Trial, Investigating the Efficacy and Safety of Repeated Lamazym Treatment of Subjects With Alpha-Mannosidosis.
Brief Title: A Placebo-Controlled Phase 3 Trial of Repeated Lamazym Treatment of Subjects With Alpha-Mannosidosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Zymenex A/S (Industry)
Collaborators: European Commission (Other)
Responsible Party: Sponsor
Organization: Chiesi Farmaceutici S.p.A. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: rhLAMAN-05; 2012-000979-17 (EudraCT Number)
Record Dates: First submitted 2012-08-22; First posted 2012-09-10 (Estimated); Last update posted 2020-08-03 (Actual); Status verified 2020-07

CONDITIONS: Alpha-Mannosidosis
MeSH Terms: conditions — alpha-Mannosidosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lamazym (Active Comparator): 1 mg Lamazym/kg body weight
  Interventions: Drug: Lamazym
- Placebo (Placebo Comparator): Placebo is formulated as an isotonic phosphate buffer with glycine and mannitol
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lamazym — ERT, i.v. infusions weekly
  Other Names: rhLAMAN; recombinant human alpha-mannosidase
  Arms: Lamazym
Drug: Placebo — Infusions weekly
  Arms: Placebo

SUMMARY:
The overall objective of this trial is to evaluate the efficacy and safety of repeated Lamazym i.v. treatment, compared with placebo, in subjects 5-35 years of age with alpha-Mannosidosis

ELIGIBILITY:
Inclusion Criteria:

* Subject or subjects legally authorized guardian(s) must provide signed, informed consent prior to performing any trial-related activities
* The subject and his/her guardian(s) must have the ability to comply with the protocol
* The subject must have a confirmed diagnosis of alpha-Mannosidosis as defined by alpha-Mannosidase activity < 10% of normal activity (historical data)
* The subject must have an age at the time of screening ≥ 5 years and ≤ 35 years
* The subject must have the ability to physically and mentally cooperate in the tests
* The subject must have an ECHO without abnormalities that, in the opinion of the Investigator, would preclude participation in the trial

Exclusion Criteria:

* The subjects diagnosis cannot be confirmed by alpha-Mannosidase activity < 10% of normal activity
* The subject cannot walk without support
* Presence of known chromosomal abnormality and syndromes affecting psychomotor development, other than alpha-Mannosidosis
* History of BMT
* Presence of known clinically significant cardiovascular, hepatic, pulmonary, or renal disease or other medical conditions that, in the opinion of the Investigator, would preclude participation in the trial
* Any other medical condition or serious intercurrent illness, or extenuating circumstance that, in the opinion of the Investigator, would preclude participation in the trial
* Pregnancy: Pregnant woman is excluded. Before start of the treatment the investigators will for women of childbearing potential perform a pregnancy test and decide whether or not there is a need for contraception
* Psychosis; any psychotic disease, also in remission, is an exclusion criteria
* Planned major surgery that, in the opinion of the Investigator, would preclude participation in the trial
* Participation in other interventional trials testing IMP (including Lamazym) within the last 3 months
* Adult patients who, in the opinion of the Investigator, would be unable to give consent, and who does not have any legal protection or guardianship
* Total IgE >800 IU/ml
* Known allergy to the IMP or any excipients (Sodium-Phosphate, Glycine, Mannitol)

Ages: 5 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Actual)
Dates: Start 2012-08; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Reduction of oligosaccharides in serum | Baseline evaluation prior to first dose, midterm evaluation after 26 weeks, and end evaluation after 52 weeks
  Primary efficacy endpoint evaluated as change from baseline in the active group versus the placebo group
The number of steps climbed in 3 minutes (3-minute stair climb test) | Baseline evaluation prior to first dose, midterm evaluation after 26 weeks, and end evaluation after 52 weeks
  Primary efficacy endpoint evaluated as change from baseline in the active group versus the placebo group

SECONDARY OUTCOMES:
Forced Vital Capacity | Baseline evaluation prior to first dose, midterm evaluation after 26 weeks, and end evaluation after 52 weeks
  Secondary efficacy endpoint evaluated as change from baseline in the active group versus the placebo group
The distance walked in 6 minutes (6-minute walk test) | Baseline evaluation prior to first dose, midterm evaluation after 26 weeks, and end evaluation after 52 weeks
  Secondary efficacy endpoint evaluated as change from baseline in the active group versus the placebo group
Adverse Events | 1 week
  Safety endpoint assessed weekly throughout the trial
Development of clinically significant changes in vital signs and change in physical examination | 1 week
  Safety endpoints assessed weekly throughout the trial
Clinical laboratory parameters (hematology, biochemistry and urinalysis) | 1 week
  Safety endpoints assessed weekly throughout the trial
Development of Lamazym antibodies and neutralizing/inhibitory antibodies | 1 week
  Safety endpoints assessed weekly throughout the trial

OTHER OUTCOMES:
Quantitative determination of rhLAMAN in plasma | 10 min, 60 min, 2 hours, 24 hours, 3 days, 7 days
  Pharmacokinetic (PK) assessments. Blood samples are drawn pre-treatment and at various times post-treatment (see time frame above)

CONTACTS AND LOCATIONS:
Overall Officials: Allan M Lund, MD, Principal Investigator — Copenhagen University Hospital, Center for Metabolic Diseases, Department for Clinical Genetics; Jens Fogh, Study Chair — Zymenex A/S
Locations (6):
- Center for Metabolic Diseases, Department of Clinical Genetics, Juliane Marie Centre, Copenhagen University Hospital, Blegdamsvej 9, Copenhagen, Denmark
- France (2):
  - Hôpital Femme Mère Enfant, Lyon, 59 boulevard Pinel, Bron
  - Hôpital Trousseau, Service de neuropédiatrie, Centre Référence des Maladies Lysosomales, 26 avenue du Docteur Arnold Netter, Paris
- Universitätsmedizin Mainz, Zentrum für Kinder- und Jugendmedizin, Langenbeckstrasse 1, Mainz, Germany
- The Children's Memorial Health Institute Warsaw, Department of Metabolic Diseases, Al Dzieci Polskich 20, Warsaw, Poland
- Genetic Medicine, 6th floor, St Mary's Hospital, Oxford Road,, Manchester, United Kingdom

REFERENCES:
- [Background] Borgwardt L, Stensland HM, Olsen KJ, Wibrand F, Klenow HB, Beck M, Amraoui Y, Arash L, Fogh J, Nilssen O, Dali CI, Lund AM. Alpha-mannosidosis: correlation between phenotype, genotype and mutant MAN2B1 subcellular localisation. Orphanet J Rare Dis. 2015 Jun 6;10:70. doi: 10.1186/s13023-015-0286-x. PMID 26048034
- [Background] Borgwardt L, Thuesen AM, Olsen KJ, Fogh J, Dali CI, Lund AM. Cognitive profile and activities of daily living: 35 patients with alpha-mannosidosis. J Inherit Metab Dis. 2015 Nov;38(6):1119-27. doi: 10.1007/s10545-015-9862-4. Epub 2015 May 28. PMID 26016802
- [Background] Harmatz P, Cattaneo F, Ardigo D, Geraci S, Hennermann JB, Guffon N, Lund A, Hendriksz CJ, Borgwardt L. Enzyme replacement therapy with velmanase alfa (human recombinant alpha-mannosidase): Novel global treatment response model and outcomes in patients with alpha-mannosidosis. Mol Genet Metab. 2018 Jun;124(2):152-160. doi: 10.1016/j.ymgme.2018.04.003. Epub 2018 Apr 18. PMID 29716835
- [Result] Borgwardt L, Guffon N, Amraoui Y, Dali CI, De Meirleir L, Gil-Campos M, Heron B, Geraci S, Ardigo D, Cattaneo F, Fogh J, Van den Hout JMH, Beck M, Jones SA, Tylki-Szymanska A, Haugsted U, Lund AM. Efficacy and safety of Velmanase alfa in the treatment of patients with alpha-mannosidosis: results from the core and extension phase analysis of a phase III multicentre, double-blind, randomised, placebo-controlled trial. J Inherit Metab Dis. 2018 Nov;41(6):1215-1223. doi: 10.1007/s10545-018-0185-0. Epub 2018 May 30. PMID 29846843
- See also: Study Record on EU Clinical Trials Register including results — https://www.clinicaltrialsregister.eu/ctr-search/search?query=2012-000979-17